CLINICAL TRIAL: NCT02730247
Title: A Phase II Clinical Trial of the Safety and Efficacy of the Addition of Ramucirumab to Nab-paclitaxel in Previously Treated Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Trial of the Safety and Efficacy of the Addition of Ramucirumab to Nab-paclitaxel in Previously Treated Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liza Villaruz, MD (Other)
Responsible Party: Sponsor-Investigator, Liza Villaruz, MD, Assistant Professor of Medicine, Division of Hematology Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-169
Record Dates: First submitted 2016-02-24; First posted 2016-04-06 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ramucirumab; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ramucirumab + nab-paclitaxel (Experimental): Ramucirumab will be administered through a vein in the arm as a 60 minute infusion at a dose of 8 mg/kg on days 1 and 15 of a 28-day cycle.
  The nab-paclitaxel will be administered through a vein in the arm as a 30 minute infusion at a dose of 100 mg/m2 on days 1, 8 and 15 of a 28 day cycle.
  Interventions: Drug: ramucirumab; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: ramucirumab — it is administered through a vein in the arm as a 60 minute infusion at a dose of 8 mg/kg on days 1 and 15 of a 28-day cycle.
  Other Names: Cyramza
Drug: nab-paclitaxel — it is administered through a vein in the arm as a 30 minute infusion at a dose of 100 mg/m2 on days 1, 8 and 15 of a 28 day cycle.
  Other Names: Abraxane

SUMMARY:
The subjects who take part in this clinical research study have advanced non-small cell lung cancer (NSCLC) that has been previously treated with other drugs. If they join this study, they would receive ramucirumab (Cyramza ®) in combination with nab-paclitaxel (Abraxane®). Ramucirumab given with nab-paclitaxel is considered an investigational drug combination to use in this type of cancer because giving these two drugs together has not been approved by any regulatory authority like the US Food and Drug Administration (FDA) for NSCLC cancer. Ramucirumab works by slowing or stopping the growth of cancer cells. Nab-Paclitaxel works by blocking the ability of cancer cells to break down the internal 'skeleton' that allows them to divide and multiply. With the skeleton still in place, the cells cannot divide and they eventually die.

DETAILED DESCRIPTION:
Ramucirumab is a human IgG1 (Immunoglobulin G) monoclonal antibody that targets the extracellular domain of VEGFR-2 (vascular endothelial growth factor receptor). A recent double-blind, placebo-controlled clinical trial evaluated the addition of ramucirumab to docetaxel compared with docetaxel and placebo in patients with Stage IV squamous and non-squamous NSCLC in the 2nd-line treatment setting. This study demonstrated a superior overall survival (OS), progression-free survival (PFS), and overall response rate (ORR) with the combination therapy compared with docetaxel with placebo. This effect was seen across histologic subtypes, in the absence of excess toxicity in patients with squamous cell histology. This finding is intriguing, as prior study of bevacizumab in patients with NSCLC of squamous cell histology was associated with excess pulmonary hemorrhage. This provides the rationale for further investigation of ramucirumab in patients with squamous cell NSCLC.

nab-Paclitaxel is a formulation of paclitaxel complexed with albumin that is readily soluble in saline and allows administration of paclitaxel without the use of lipid-based solvents and the need for corticosteroid and antihistamine premedication. nab-Paclitaxel was approved for the 1st line treatment of NSCLC based on a trial which demonstrated a superior ORR with the addition of nab-paclitaxel to carboplatin compared with carboplatin/paclitaxel in patients with advanced and metastatic NSCLC, as well as prolonged PFS and OS without statistical significance. The subgroup analysis by tumor histology demonstrated a statistically significant advantage for nab-paclitaxel/carboplatin in terms of best overall response rate (41% vs 24%, p<0.001), and numerically better PFS and OS in squamous NSCLC. [3]

This is a single-arm phase II clinical trial, in which patients with previously treated NSCLC will be treated with ramucirumab/nab-paclitaxel until disease progression, unacceptable treatment-related toxicity or withdrawal of consent with the primary endpoint of progression-free survival. A minimum of 40 patients with squamous cell histology will be required for determination of the co-primary endpoint. The investigators hypothesize that the addition of ramucirumab to nab-paclitaxel is well-tolerated and associated with a superior PFS compared with single agent taxane-based therapy.

ELIGIBILITY:
Inclusion Criteria:

All patients must have or meet the following:

* Histologically or cytologically confirmed Stage IV (AJCC 7) non-small cell lung cancer.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Received at least one prior platinum-based chemotherapy for locally advanced or metastatic disease. Prior bevacizumab as 1st line and/or maintenance therapy is allowed. Prior nivolumab is allowed.
* Age ≥18 years.
* ECOG performance status ≤2
* Life expectancy of greater than 12 weeks.
* Adequate liver function
* Adequate hematologic function
* Not have cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) with a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
* Adequate renal function
* Urinary protein of ≤1+ on dipstick or routine urinalysis (UA).
* Adequate coagulation function. Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy.
* Treated and clinically stable brain metastases are allowed.
* Adequate contraceptive use.
* < Grade 2 pre-existing peripheral neuropathy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with previous intolerance to ramucirumab.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ramucirumab or nab-paclitaxel.
* Patients with untreated CNS metastases.
* Patients with significant bleeding disorders, vasculitis, or who experienced Grade 3/4 gastrointestinal (GI) bleeding within 3 months prior to enrollment.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to enrollment.
* Any arterial thromboembolic events, within 6 months prior to enrollment.
* History of uncontrolled hereditary or acquired thrombotic disorder.
* Uncontrolled or poorly-controlled hypertension.
* A serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment.
* Chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Elective or planned major surgery scheduled during the course of the clinical trial.
* Hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon) within 2 months prior to enrollment, or with central or cavitating lesions.
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* History of GI perforation and/or fistulae within 6 months prior to enrollment, or risk factors for perforation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy
* HIV-positive patients on combination antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2019-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Villaruz, MD, Principal Investigator — University of Pittsburgh Cancer Institute, Department of Hematology Oncology
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab + Nab-paclitaxel: 8 mg/kg IV ramucirumab on days 1 and 15 of a 28-day treatment cycle
  100 mg/m^2 IV nab-paclitaxel on days 1, 8 and 15 of a 28 day cycle
Period: Overall Study
Arm/Group | Ramucirumab + Nab-paclitaxel
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 63 [54.9 to 77.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Stage of Disease [Count of Participants; unit: Participants] — Stage IV and Stage IV B: Cancer has spread to other body organs (metastasis); possibly including lymph nodes.
  Participants
    Stage IV | 5
    Stage IV B | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Grade 2: In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    Grade 1 | 6
    Grade 2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The duration of time from start of treatment to time of progression or death. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 26 months
Population: Patients evaluable for clinical response who have received at least one cycle of therapy.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
months | 8.16 [3.68 to NA] — Upper bound not able to be reached due to low patient accrual.

2. Primary Outcome: Worst Grade of Adverse Event Experienced
Description: Percentage of patients that experienced Grade 3-5 adverse events as their highest Grade event, irrespective of relatedness to treatment, per NCI CTCAE v2.0 (National Cancer Institute Common Terminology Criteria for Adverse Events).
Time Frame: Up to 26 months
Population: Patients that received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
percentage of participants
  Grade 3 adverse event | 57.1 [20.0 to 87.6]
  Grade 4 adverse event | 28.6 [6.2 to 70.7]
  Grade 5 adverse event | 14.3 [1.8 to 59.7]

3. Primary Outcome: Worst Grade of Adverse Event Experienced, at Least Possibly Related to Treatment
Description: Percentage of patients who experienced Grade 2-5 adverse events as their highest Grade event, that were at least possibly related to treatment, per NCI CTCAE v2.0 (National Cancer Institute Common Terminology Criteria for Adverse Events).
Time Frame: Up to 26 months
Population: Patients that received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
percentage of participants
  Grade 2 | 14.3 [1.5 to 64.8]
  Grade 3 | 42.9 [10.5 to 82.8]
  Grade 4 | 28.6 [5.2 to 74.6]
  Grade 5 | 14.3 [1.5 to 64.8]

4. Primary Outcome: Worst Grade of Adverse Event Experienced, at Least Probably Related to Treatment
Description: Percentage of patients who experienced Grade 0-4 adverse events as their highest Grade event, that were at least probably related to treatment, per NCI CTCAE v2.0 (National Cancer Institute Common Terminology Criteria for Adverse Events).
Time Frame: Up to 26 months
Population: Patients that received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
percentage of participants
  Grade 0 | 14.3 [1.3 to 68.4]
  Grade 1 | 28.6 [4.5 to 77.3]
  Grade 2 | 28.6 [4.5 to 77.3]
  Grade 3 | 14.3 [1.3 to 68.4]
  Grade 4 | 14.3 [1.3 to 68.4]

5. Primary Outcome: Worst Grade of Adverse Event Experienced, Definitely Related to Treatment
Description: Percentage of patients that experienced Grade 0-2 adverse events as their highest Grade event, that were definitely related to treatment, per NCI CTCAE v2.0 (National Cancer Institute Common Terminology Criteria for Adverse Events.
Time Frame: Up to 26 months
Population: Patients that received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
proportion of participants
  Grade 0 | 71.4 [29.3 to 93.8]
  Grade 1 | 14.3 [1.8 to 59.7]
  Grade 2 | 14.3 [1.8 to 59.7]

6. Secondary Outcome: Best Overall Response
Description: Median percentage of patients who experienced a best response of partial or complete response (PR + CR) / total number of patients (PR + CR + Stable Disease (SD) + Progressive Disease (PD)), per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm; appearance new lesions.
Time Frame: Up to 26 months
Population: Patients evaluable for response who received at least one cycle of therapy.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 6
percentage of participants
  Best Response - Stable Disease | 67.7 [22.3 to 95.7]
  Best Response - Partial Response | 33.3 [4.3 to 77.8]

7. Secondary Outcome: Overall Survival (OS)
Description: The duration of time from the start of treatment to death.
Time Frame: Up to 26 months
Population: All enrolled participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
months | 7.42 [3.48 to NA] — Upper bound not able to be reached due to low patient accrual.

8. Secondary Outcome: Median EuroQol Five Dimension Questionnaire (EQ-5D-5L) Score
Description: The EuroQol Five Dimension questionnaire (EQ-5D-5L) score is a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: level 0=no problems, level 1=slight problems, level 2=moderate problems, level 3=severe problems and level 4= extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  Data is presented as a health profile table reporting a proportion of reported problems for each level for each dimension and/or dichotomised levels - 'no problems' (i.e. level 1) and 'problems' (i.e. levels 2 to 5)
Time Frame: Baseline through up to 26 months
Population: Patients that received at least one dose of study treatment and who completed at least one questionnaire.
Measure: Median (Full Range); unit: EQ-5D-5L score
Arm/Group | Ramucirumab + Nab-paclitaxel
Number analyzed (Participants) | 7
EQ-5D-5L score
  Walking | 1 [0 to 2]
  Dressing | 1 [0 to 2]
  Active | 1 [0 to 4]
  Pain | 1 [0 to 4]
  Anxious | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: Up to 26 months
Arm/Group | Ramucirumab + Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Nab-paclitaxel (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Cardiac arrest (Cardiac disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (8)
Lymphocyte count decreased (Investigations) | 3 (16)
Neutrophil count decreased (Investigations) | 3 (24)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (2)
Weight loss (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 2 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Nab-paclitaxel (N=7)
Alkaline phosphatase increased (Investigations) | 3 (14)
Anemia (Blood and lymphatic system disorders) | 6 (56)
Anorexia (Metabolism and nutrition disorders) | 4 (8)
Anxiety (Psychiatric disorders) | 1 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 3 (20)
Blood bilirubin increased (Investigations) | 2 (14)
Cardiac arrest (Cardiac disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Creatinine increased (Investigations) | 1 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (4)
Depression (Psychiatric disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (8)
Dysgeusia (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Edema limbs (General disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (2)
Fatigue (General disorders) | 5 (16)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Gait disturbance (General disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (30)
Hypertension (Vascular disorders) | 2 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (48)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (36)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (14)
Hypotension (Vascular disorders) | 1 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
INR increased (Investigations) | 1 (4)
Investigations - Other, specify (Investigations) | 3 (14)
Lymphocyte count decreased (Investigations) | 3 (30)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (10)
Mucosal infection (Infections and infestations) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Neutrophil count decreased (Investigations) | 5 (84)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Platelet count decreased (Investigations) | 3 (22)
Proteinuria (Renal and urinary disorders) | 4 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 2 (8)
Skin infection (Infections and infestations) | 2 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4)
Upper respiratory infection (Infections and infestations) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Weight loss (Investigations) | 2 (6)
White blood cell decreased (Investigations) | 4 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02730247/Prot_SAP_000.pdf